CLINICAL TRIAL: NCT06106074
Title: A Randomized, Double-blind, Placebo-controlled Study of the Tolerability and Pharmacokinetics of Ascending Single and 14-day Repeated Oral Doses of SAR442168 With a Food Effect Investigation in Healthy Adult Participants
Brief Title: Study of the Tolerability and Pharmacokinetics of Oral Doses of SAR442168 With a Food Effect Investigation in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TDU16831-TDR16862
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1a (Experimental): 3 single ascending doses of SAR442168 or placebo in fasted and fed (high-fat breakfast) conditions
  Interventions: Drug: Tolebrutinib; Drug: Placebo
- Part 1b (Experimental): 2 single doses of SAR442168 under fed conditions (moderate-fat breakfast).
  Interventions: Drug: Tolebrutinib
- Part 1c (Experimental): 1 single dose of SAR442168 under fasting and fed conditions (high-fat breakfast).
  Interventions: Drug: Tolebrutinib
- Part 1d (Experimental): 1 single dose of SAR442168 under fasting and fed conditions (Standardized high-fat breakfast).
  Interventions: Drug: Tolebrutinib
- Part 2 (Experimental): 3 ascending once-daily repeated single doses of SAR442168 or placebo for 14 days under fed conditions (moderate-fat breakfast)
  Interventions: Drug: Tolebrutinib; Drug: Placebo

INTERVENTIONS:
Drug: Tolebrutinib — Tablet, oral
  Other Names: SAR442168
Drug: Placebo — Tablet, oral
  Arms: Part 1a; Part 2

SUMMARY:
This is a randomized, placebo-controlled, four-part, Phase I, first in human (FIH) study to assess the tolerability and pharmacokinetics (PK) of ascending single and 14-day repeated oral doses of SAR442168 with a food effect investigation in healthy adult participants.

* In Part 1a: The tolerability and safety of SAR442168 and the pharmacokinetic parameters of SAR442168 and metabolite(s)after ascending single oral doses in fasted and fed conditions
* In Part 1b: The relationship of PK of SAR442168 and metabolite(s) in cerebrospinal fluid (CSF) to that in plasma after single oral doses given in fed conditions (moderate-fat meal)
* In Part 1c: The effect of a high-fat meal on the pharmacokinetics of SAR442168 and metabolite(s) (high-fat)
* In Part 1d: The effect of a high-fat meal on the pharmacokinetics of SAR442168 and metabolite(s) (standardized high-fat meal)
* In Part 2: The tolerability and safety of SAR442168 and the pharmacokinetic parameters of SAR442168 and metabolite(s) after 14-day ascending repeated oral doses of SAR442168 given in fed conditions (moderate-fat meal).

ELIGIBILITY:
Inclusion Criteria:

* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Part 1a and Part 2: Number of participants with Adverse Events (AEs) and treatment-emergent adverse events (TEAEs) | Part 1a: Day 1 to approximately Day 14 Part 2: Day 1 to approximately Day 21
Part 1b: Total (free and bound) SAR442168 concentrations in CSF | From Day 1 to Day 3
Part 1b: Total (free and bound) SAR442168 metabolite(s) concentrations in CSF | From Day 1 to Day 3
Part 1c and Part 1d: Maximum plasma concentration observed (Cmax) ratio fed/fast of SAR442168 | From Day 1 to Day approximately 14
Part 1c and Part1d: Cmax ratio fed/fasted of SAR442168 metabolite(s) | From Day 1 to Day approximately 14
Part 1c and Part 1d: Area under the plasma concentration versus time curve (AUC) ratio fed/fast of SAR442168 | From Day 1 to Day approximately 14
Part 1c and Part1d: AUC ratio fed/fast of SAR442168 metabolite(s) | From Day 1 to Day approximately 14

SECONDARY OUTCOMES:
All Parts: Cmax of SAR442168 | From Day 1 to Day approximately 14
All Parts: Cmax of SAR442168 metabolite(s) | From Day 1 to Day approximately 14
Part 1a, Part 1b and Part 2: tmax of SAR442168 | From Day 1 to Day approximately 14
Part 1a, Part 1b and Part 2: tmax of SAR442168 metabolite(s) | From Day 1 to Day approximately 14
Part 1a, Part 1b, Part1c and Part 1d: AUC of SAR442168 | From Day 1 to Day approximately 14
Part 1a, Part 1b, Part1c and Part 1d: AUC of SAR442168 metabolite(s) | From Day 1 to Day approximately 14
Part 2: AUC0-tau for SAR442168 | From Day 1 to Day approximately 14
  Area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (24 hours)
Part 2: AUC0-tau for SAR442168 metabolite(s) | From Day 1 to Day approximately 14
  Area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (24 hours)
Part 1b, Part1c and 1d: Number of participants with Adverse Events (AEs) and treatment-emergent adverse events (TEAEs) | From Day 1 to Day approximately 14

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- New Orleans Clinical Research Site Number : 8400001, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org